CLINICAL TRIAL: NCT07227428
Title: Comparison of Glucocorticoid Tapering Schedules in Rheumatoid Arthritis.
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); SMG-SNU Boramae Medical Center (Other); Gachon University Gil Medical Center (Other); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Responsible Party: Principal Investigator, Eun Bong Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2502-080-1613
Record Dates: First submitted 2025-11-07; First posted 2025-11-12 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: steroid taper; adrenal insufficiency; disease activity
MeSH Terms: conditions — Arthritis, Rheumatoid; Adrenal Insufficiency | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This study is a single-blind study without placebo control. Investigators who access the DAS28 will be blinded to the treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 5mg tablet taper (Experimental): Prednisolone will be tapered using 5mg tablet formulation
  Interventions: Drug: Prednisolone
- 1mg tablet taper (Active Comparator): Prednisolone will be tapered using 1 mg tablet formulation
  Interventions: Drug: Prednisolone
- Continue (Placebo Comparator): Prednisolone will be continued
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Prednisolone — PD will be tapered using a 5mg tab formulation
  Arms: 5mg tablet taper
Drug: Prednisolone — PD will be tapered using a 1 mg tab formulation
  Arms: 1mg tablet taper
Drug: Prednisolone — PD will be continued
  Arms: Continue

SUMMARY:
This multicenter, randomized, controlled, single-blind prospective study aims to establish an evidence-based protocol for discontinuing long-term low-dose glucocorticoids in patients with rheumatoid arthritis (RA). The study will compare two tapering strategies (1) a split-dose tapering method, in which the 5 mg tablet is divided into halves and gradually reduced, and (2) a sequential 1 mg-by-1 mg tapering method.

A total of 206 patients (including 50 from Seoul National University Hospital) will be enrolled and followed for six months. Participants will be randomly assigned to one of the two tapering arms, and an exploratory group will include patients who continue low-dose prednisolone without tapering.

The primary efficacy endpoint is the change in RA disease activity, measured by DAS28-CRP, to demonstrate non-inferiority between the two tapering strategies. Secondary endpoints include the success rate of glucocorticoid discontinuation and changes in disease activity over time.

This trial seeks to define a standardized, practical glucocorticoid tapering protocol tailored to Korean RA patients. The findings are expected to support safer steroid withdrawal, reduce treatment-related adverse events, and guide clinical decision-making in long-term management of rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥19 years of age at time of consent
* Body weight < 90kg
* Have a diagnosis of RA per the 2010 ACR/EULAR criteria for at least 6 months
* Disease activity of rheumatoid arthritis has been stable for at least 4 weeks prior to randomization (DAS28-CRP ≤ 3.2)
* The patient has been taking a stable dose of prednisolone equivalent ≤ 5 mg/day for at least 12 weeks prior to randomization
* The dose of corticosteroids has not changed during the 4 weeks prior to randomization

Exclusion Criteria:

* History of major surgery within 8 weeks prior to screening
* Increase in the dose of antirheumatic drugs within 4 weeks prior to screening due to worsening arthritis
* Pregnant or breastfeeding
* RA functional class IV, requiring confinement to bed or wheelchair
* History of primary or secondary adrenal insufficiency

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease Activity Score 28-CRP | 6 months
  Disease activity: Remission <2.6; Low 2.6-3.2; Moderate >3.2-5.1 High >5.1

SECONDARY OUTCOMES:
Number of Participants with RA flare | 6 months
Number of adrenal insufficiency | 6 months
Frequency of rescue medication use (%) | 6 months
Rate of successful steroid discontinuation (%) | 6 months

IPD SHARING:
Plan to Share IPD: Undecided